CLINICAL TRIAL: NCT06091371
Title: Prospective Evaluation of Patients Undergoing Surgical Treatment for Arthrorisis of the Subtalar Joint With a Polymeric Endorthesis for the Treatment of Flexible Flatfoot in the Growth Age
Brief Title: Arthrorisis of the Subtalar Joint With a Polymeric Endorthesis for Flexible Flatfoot Treatment During the Growth Age Prospective Evaluation
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Antonio Mazzotti, Principal Investigator, Istituto Ortopedico Rizzoli
Other Study IDs: EPProsp
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Subtalar Arthrorisis; Flat Feet; Growth Age
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Arthrorisis of the subastragalus joint represents one of the surgical treatments for addressing flexible flatfoot, a condition caused by joint deformity. The device is designed to restore the correct joint relationships between the astragalus and calcaneus, with the goal of maintaining the new and proper joint alignment over time, typically allowing for bone remodeling along natural growth lines, usually within a few years.

Several implants and various variations of the procedure have been developed.There are currently no prospective studies that assess radiographic and clinical data over time. Therefore, the purpose of this study is to prospectively analyze the outcomes of surgical intervention using subastragalus arthrorisis with a polymeric endorthesis for the treatment of flexible flatfoot during the growth period in a consecutive series of 55 patients.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic, flexible, symptomatic flatfoot
* Patients aged between 8 and 14 years

Exclusion Criteria:

* Joint laxity
* Neuromuscular disorders
* Neurological conditions
* Traumatic sequelae
* Iatrogenic flatfoot
* Congenital flatfoot due to tarsal synostosis

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients aged between 8 and 14 years with idiopathic, flexible, symptomatic flatfoot
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Meary's angle | At baseline (day 0)
  Meary's angle is the angle between a line drawn along the longitudinal axes of the talus (mid-talar axis) and the first metatarsal (first metatarsal axis) on the lateral weight bearing X ray.
Meary's angle | After 1 month
  Meary's angle is the angle between a line drawn along the longitudinal axes of the talus (mid-talar axis) and the first metatarsal (first metatarsal axis) on the lateral weight bearing X ray.
Meary's angle | After 3 months
  Meary's angle is the angle between a line drawn along the longitudinal axes of the talus (mid-talar axis) and the first metatarsal (first metatarsal axis) on the lateral weight bearing X ray.
Meary's angle | After 6 months
  Meary's angle is the angle between a line drawn along the longitudinal axes of the talus (mid-talar axis) and the first metatarsal (first metatarsal axis) on the lateral weight bearing X ray.
Meary's angle | After 12 months
  Meary's angle is the angle between a line drawn along the longitudinal axes of the talus (mid-talar axis) and the first metatarsal (first metatarsal axis) on the lateral weight bearing X ray.
Meary's angle | After 24 months
  Meary's angle is the angle between a line drawn along the longitudinal axes of the talus (mid-talar axis) and the first metatarsal (first metatarsal axis) on the lateral weight bearing X ray.
Meary's angle | After 36 months
  Meary's angle is the angle between a line drawn along the longitudinal axes of the talus (mid-talar axis) and the first metatarsal (first metatarsal axis) on the lateral weight bearing X ray.
Meary's angle | After 48 months
  Meary's angle is the angle between a line drawn along the longitudinal axes of the talus (mid-talar axis) and the first metatarsal (first metatarsal axis) on the lateral weight bearing X ray.
Meary's angle | After 72 months
  Meary's angle is the angle between a line drawn along the longitudinal axes of the talus (mid-talar axis) and the first metatarsal (first metatarsal axis) on the lateral weight bearing X ray.

SECONDARY OUTCOMES:
AOFAS Score | At baseline (day 0)
  The American Orthopedic Foot and Ankle Society Score is a semi-objective rating scale that evaluates ankle pain, motion and alignment and ranges from 0 to 100 points. 0 worst possible score, 100 best possible score
AOFAS Score | After 1 month
  The American Orthopedic Foot and Ankle Society Score is a semi-objective rating scale that evaluates ankle pain, motion and alignment and ranges from 0 to 100 points. 0 worst possible score, 100 best possible score
AOFAS Score | After 3 months
  The American Orthopedic Foot and Ankle Society Score is a semi-objective rating scale that evaluates ankle pain, motion and alignment and ranges from 0 to 100 points. 0 worst possible score, 100 best possible score
AOFAS Score | After 6 months
  The American Orthopedic Foot and Ankle Society Score is a semi-objective rating scale that evaluates ankle pain, motion and alignment and ranges from 0 to 100 points. 0 worst possible score, 100 best possible score
AOFAS Score | After 12 months
  American Orthopaedic Foot and Ankle Society Score- from 0 to 100 points. 0 worst possible score, 100 best possible score
AOFAS Score | After 24 months
  American Orthopaedic Foot and Ankle Society Score- from 0 to 100 points. 0 worst possible score, 100 best possible score
AOFAS Score | After 36 months
  American Orthopaedic Foot and Ankle Society Score- from 0 to 100 points. 0 worst possible score, 100 best possible score
AOFAS Score | After 48 months
  American Orthopaedic Foot and Ankle Society Score- from 0 to 100 points. 0 worst possible score, 100 best possible score
AOFAS Score | After 72 months
  American Orthopaedic Foot and Ankle Society Score- from 0 to 100 points. 0 worst possible score, 100 best possible score

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nelson SC, Haycock DM, Little ER. Flexible flatfoot treatment with arthroereisis: radiographic improvement and child health survey analysis. J Foot Ankle Surg. 2004 May-Jun;43(3):144-55. doi: 10.1053/j.jfas.2004.03.012. PMID 15181430